CLINICAL TRIAL: NCT05956587
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of SI-B003 Monotherapy and BL-B01D1+SI-B003 Combination Therapy in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer, Nasopharyngeal Carcinoma and Other Solid Tumors
Brief Title: A Study of SI-B003 and BL-B01D1+SI-B003 in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer, Nasopharyngeal Carcinoma and Other Solid Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-SI-B003-201-01
Record Dates: First submitted 2023-07-13; First posted 2023-07-21 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Non-small Cell Lung Cancer; Nasopharyngeal Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study treatment (Experimental): Participants received SI-B003 and BL-B01D1+SI-B003 in the first cycle (3 weeks). Participants who had a clinical benefit could receive additional cycles of additional treatment. Administration will be discontinued because of disease progression or intolerable toxicity or for other reasons.
  Interventions: Drug: BL-B01D1; Drug: SI-B003

INTERVENTIONS:
Drug: BL-B01D1 — Administration by intravenous infusion
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
Drug: SI-B003 — Administration by intravenous infusion

SUMMARY:
Phase II: To explore the efficacy, safety and tolerability of BL-B01D1+SI-B003 in patients with locally advanced or metastatic non-small cell lung cancer and nasopharyngeal carcinoma, and to further explore the optimal dose and mode of combination.

DETAILED DESCRIPTION:
Phase II: To explore the efficacy of BL-B01D1+SI-B003 combination in patients with locally advanced or metastatic solid tumors such as non-small cell lung cancer and nasopharyngeal carcinoma. To explore the safety and tolerability of BL-B01D1+SI-B003 combination in patients with locally advanced or metastatic non-small cell lung cancer and nasopharyngeal carcinoma, and to further explore the optimal dose and mode of combination.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form voluntarily and follow the protocol requirements;
2. Gender is not limited;
3. Age: ≥18 years old and ≤75 years old;
4. Expected survival time ≥3 months;
5. Patients with histologically and/or cytologically confirmed locally advanced or metastatic solid tumors such as non-small cell lung cancer and nasopharyngeal carcinoma;
6. Consent to provide archival tumor tissue samples or fresh tissue samples from primary or metastatic lesions within 2 years;
7. At least one measurable lesion meeting the RECIST v1.1 definition was required;
8. ECOG 0 or 1;
9. The toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0;
10. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
11. No blood transfusion, no use of cell growth factors and/or platelet raising drugs within 14 days before the first use of the study drug, and the level of organ function must meet the requirements;
12. Coagulation function: international normalized ratio ≤1.5, and activated partial thromboplastin time≤1.5 ULN;
13. Urinary protein ≤2+ or ≤1000mg/24h;
14. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before starting treatment, serum or urine must be negative for pregnancy, and must be non-lactating; All enrolled patients (male or female) were advised to use adequate barrier contraception throughout the treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. For stage 3 Cohort_A, patients with MET 14 exon skipping detected by gene sequencing report before signing informed consent;
2. Chemotherapy, biological therapy and other anti-tumor therapies have been used within 4 weeks or 5 half-lives before the first dose; Mitomycin and nitrosoureas were administered within 6 weeks before the first dose; Oral drugs such as fluorouracil;
3. Had received immunotherapy and developed ≥ grade 3 irAE or ≥ grade 2 immune-related myocarditis;
4. Use of immunomodulatory drugs within 14 days before the first dose of study drug;
5. History of severe heart disease;
6. QT prolongation, complete left bundle branch block, III degree atrioventricular block;
7. Systemic corticosteroids or immunosuppressive agents are required within 2 weeks before study dosing;
8. Active autoimmune and inflammatory diseases;
9. Other malignancies diagnosed within 5 years before the first dose;
10. Hypertension poorly controlled by two antihypertensive drugs;
11. Pulmonary disease was defined as grade ≥3 according to CTCAE v5.0; Patients with current or history of ILD;
12. Unstable thrombotic events requiring therapeutic intervention within 6 months before screening;
13. Patients with a large amount of serous cavity effusion, or serous cavity effusion with symptoms, or within 4 weeks before signing informed consent;
14. Patients with active central nervous system metastases;
15. Patients with a history of allergy to recombinant humanized antibody or human-mouse chimeric antibody or to any excipients of the test drug;
16. Prior organ transplantation or allogeneic hematopoietic stem cell transplantation;
17. Human immunodeficiency virus antibody positive, active tuberculosis, active hepatitis B virus infection or hepatitis C virus infection;
18. Active infection requiring systemic therapy;
19. Had participated in another clinical trial within 4 weeks before the first dose;
20. The investigator did not consider it appropriate to use other conditions for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study of SI-B003.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the first dose of medication to disease progression or death, whichever occurred first.
Disease control rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any adverse and unexpected change in body structure, function, or chemistry or any exacerbation of an existing condition (i.e., any clinically significant adverse change in frequency and/or intensity) during treatment. The type, frequency, and severity of TEAE will be assessed during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, PHD, Principal Investigator — Sun Yat-sen University
Locations (16):
- China (16):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital Tongji Medical College， Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Hunan Cancer Hospita, Changsha, Hunan
  - The Second Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - Linyi Cancer Hospital, Linyi, Shangdong
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi’an, Shanxi
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang